CLINICAL TRIAL: NCT01640964
Title: An Exploratory Study to Investigate the Haemodynamic Effects of Serelaxin (RLX030) in Patients With Compensated Cirrhosis and Portal Hypertension
Brief Title: An Exploratory Haemodynamic Study in Patients With Compensated Cirrhosis and Portal Hypertension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRLX030X2201; 2012-000236-26 (EudraCT Number)
Record Dates: First submitted 2012-06-21; First posted 2012-07-16 (Estimated); Results first posted 2016-01-20 (Estimated); Last update posted 2016-03-15 (Estimated); Status verified 2016-03

CONDITIONS: Compensated Cirrhosis and Portal Hypertension
Keywords: Portal hypertension, cirrhosis, TIPSS, MRI, MRA, portal pressure, portal pressure gradient
MeSH Terms: conditions — Hypertension, Portal; Fibrosis | interventions — Terlipressin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Part A: Terlipressin acetate (Experimental): Patients received terlipressin acetate 2 mg intravenous (IV) bolus injection.
  Interventions: Drug: Terlipressin acetate
- Part A: Serelaxin (RLX030) (Experimental): Randomized patients received an intravenous serelaxin infusion at two different infusion rates: 80 μg/kg/day for 60 min followed by 30 μg/kg/day for at least 60 min.; duration of infusion depends on time required for completion of magnetic resonance angiography (MRA) data acquisition
  Interventions: Drug: Serelaxin (RLX030)
- Part B Serelaxin (RLX030) (Experimental): The patients enrolled in this part of the study received an intravenous (iv) serelaxin infusion at two different infusion rates: 80 μg/kg/day for 60 min followed by 30 μg/kg/day for at least 60 min; duration of infusion depends on time required for completion of Portal pressure gradient (PPG) data acquisition.
  Interventions: Drug: Serelaxin (RLX030)

INTERVENTIONS:
Drug: Terlipressin acetate — IV bolus injection
  Arms: Part A: Terlipressin acetate
Drug: Serelaxin (RLX030) — Part A2: IV infusion for 2-3 hours; duration of infusion depends on time required for completion of MRA data acquisition; Part B: IV infusion for approximately 2 hours
  Arms: Part A: Serelaxin (RLX030); Part B Serelaxin (RLX030)

SUMMARY:
The main purpose of this exploratory study was to investigate the effect of serelaxin (RLX030) infusion on the hepatic and renal circulation in patients with compensated cirrhosis and portal hypertension. Measurements were acquired non-invasively using magnetic resonance angiography (MRA) (study part A) and more directly via cannulation of the hepatic portal vein during a routine transjugular intrahepatic portosystemic shunt (TIPSS) check procedure (study part B), to determine the acute haemodynamic response to serelaxin (RLX030).

ELIGIBILITY:
Inclusion Criteria:

Study Parts A and B:

-Cirrhosis of alcohol aetiology according to physician's assessment prior to screening.

Part A:

-Cirrhosis with clinical and/or endoscopic evidence of portal hypertension (e.g. oesophageal varices).

Part B:

* Cirrhosis with TIPSS in situ and PPG>5mmHg.
* Fully functioning TIPSS without variceal filling as confirmed by portography.

Exclusion Criteria:

Study Parts A and B:

* Use of any drug to treat portal hypertension (e.g. vasodilators such as non-selective beta blockers or nitrates) within 1 month prior to screening.
* Decompensated cirrhosis (Child-Pugh score >9 points, and/or ascites requiring diuretics, and/or hepatic encephalopathy) at visit 1.
* Presence of any non-controlled and clinically significant disease that could affect the study outcome or that would place the patient at undue risk.

Part A:

* BMI (weight[kg] / height[m^2]) > 40 kg/m^2.
* Any contraindication to having an MRI scan

Part B:

-Contraindication to catheterization

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2013-04; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, Edinburgh, United Kingdom

REFERENCES:
- [Derived] Snowdon VK, Lachlan NJ, Hoy AM, Hadoke PW, Semple SI, Patel D, Mungall W, Kendall TJ, Thomson A, Lennen RJ, Jansen MA, Moran CM, Pellicoro A, Ramachandran P, Shaw I, Aucott RL, Severin T, Saini R, Pak J, Yates D, Dongre N, Duffield JS, Webb DJ, Iredale JP, Hayes PC, Fallowfield JA. Serelaxin as a potential treatment for renal dysfunction in cirrhosis: Preclinical evaluation and results of a randomized phase 2 trial. PLoS Med. 2017 Feb 28;14(2):e1002248. doi: 10.1371/journal.pmed.1002248. eCollection 2017 Feb. PMID 28245243

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Out of 47 enrolled patients, 1 patient did not get randomized to Part A serelaxin arm ; patient withdrew consent due to failure of meeting an exclusion criterion for Part A prior to receiving the dose of study medication.
Groups:
- Part B: Serelaxin (RLX030): The patients enrolled in this part of the study received an intravenous (iv) serelaxin infusion at two different infusion rates: 80 μg/kg/day for 60 min followed by 30 μg/kg/day for at least 60 min; duration of infusion depends on time required for completion of the Portal pressure gradient (PPG) data acquisition.
Period: Overall Study
Arm/Group | Part A: Terlipressin Acetate | Part A: Serelaxin (RLX030) | Part B: Serelaxin (RLX030)
Started | 20 | 20 | 6
Completed | 19 | 19 | 3
Not Completed | 1 | 1 | 3
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Protocol Deviation | 1 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A: Terlipressin Acetate | Part A: Serelaxin (RLX030) | Part B: Serelaxin (RLX030) | Total
Number analyzed (Participants) | 20 | 20 | 6 | 46
Age, Customized [Number; unit: Patients]
  < 65 years | 17 | 15 | 6 | 38
  >= 65 years | 3 | 5 | 0 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 3 | 11
  Male | 16 | 16 | 3 | 35

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline of the Blood Flow for the Total Renal Arteries (Study Part A (Serelaxin Treatment Group Only))
Description: The flow is the average flow over the cardiac cycle. Total renal artery flow = left renal artery flow + right renal artery flow. These measurements were collected through magnetic resonance angiography (MRA) scans. Baseline blood flow for total renal artery is measured at pre-dose (Day 1, 0 min post-treatment)
Time Frame: Baseline, 120 min post serelaxin infusion
Population: Full analysis set (FAS) included all patients who received any amount of study treatment during the treatment period and had at least one post-Baseline assessment during that period.
Measure: Mean (95% Confidence Interval); unit: L/min
Arm/Group | Part A: Serelaxin (RLX030)
Number analyzed (Participants) | 20
L/min | 0.438 [0.274 to 0.601]

2. Primary Outcome: Change From Baseline of the Portal Pressure Gradient (PPG) (Study Part B)
Description: Direct venous pressure was measured by portal pressure gradient (PPG). PPG = portal vein pressure (PVP) - inferior vena cava pressure (IVCP).
  Baseline blood flow for PPG was measured at pre-dose (Day 1, 0 min post-treatment). PVP was measured at 15 min intervals (i.e. prior to and at 15, 30, 45, 60, 75, 90, 105, and 120 min of serelaxin infusion).
Time Frame: Baseline, 120 min post-infusion start
Population: For Part B of the study, full analysis set included all patients who received any amount of study treatment during the treatment period and had at least one post-baseline assessment during that period.Only patients with a value at both baseline and this time point are included.
Measure: Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Part B: Serelaxin (RLX030)
Number analyzed (Participants) | 6
mmHg | -1.2 [-6.1 to 3.7]

3. Secondary Outcome: Change From Baseline of the Blood Flow for the Total Renal Arteries (Study Part A (Terlipressin Acetate Group Only))
Description: as for outcome 1
Time Frame: Baseline, 120 min post infusion
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: L/min
Arm/Group | Part A: Terlipressin Acetate
Number analyzed (Participants) | 19
L/min | 0.059 [-0.045 to 0.164]

4. Secondary Outcome: Change From Baseline of the Blood Flow for the Hepatic Artery (Study Part A (Serelaxin Treatment Group Only))
Description: A non-contrast magnetic resonance angiography (MRA) sequence was performed to acquire phase contrast blood flow measurements from vessels of interest such as hepatic artery. The flow is the average flow over the cardiac cycle.
  Baseline blood flow measurements are measured at pre-dose (Day 1, 0 min post-treatment).
Time Frame: Baseline, 120 min post-infusion
Population: For the part A of the study, full analysis set included all patients who received any amount of study treatment during the treatment period and had at least one post-baseline assessment during that period. Only patients with a value at both baseline and at the time point are included
Measure: Mean (95% Confidence Interval); unit: L/min
Arm/Group | Part A: Serelaxin (RLX030)
Number analyzed (Participants) | 20
L/min | 0.084 [-0.020 to 0.187]

5. Secondary Outcome: Change From Baseline of the Blood Flow for the Superior Mesenteric Artery (Study Part A (Serelaxin Treatment Group Only))
Description: A non-contrast magnetic resonance angiography (MRA) sequence was performed to acquire phase contrast blood flow measurements from vessels of interest such as superior mesenteric artery. The flow is the average flow over the cardiac cycle.
  Baseline blood flow measurements are measured at pre-dose (Day 1, 0 min post-treatment).
Time Frame: Baseline, 120 min post-infusion
Population: as for outcome 4
Measure: Mean (95% Confidence Interval); unit: L/min
Arm/Group | Part A: Serelaxin (RLX030)
Number analyzed (Participants) | 20
L/min | 0.002 [-0.087 to 0.090]

6. Secondary Outcome: Change From Baseline of the Blood Flow for the Descending Thoracic Aorta (Study Part A (Serelaxin Treatment Group Only))
Description: A non-contrast magnetic resonance angiography (MRA) sequence was performed to acquire phase contrast blood flow measurements from vessels of interest such as descending thoracic aorta. The flow is the average flow over the cardiac cycle.
  Baseline blood flow measurements are measured at pre-dose (Day 1, 0 min post-treatment).
Time Frame: Baseline, 120 min post-infusion
Population: as for outcome 4
Measure: Mean (95% Confidence Interval); unit: L/min
Arm/Group | Part A: Serelaxin (RLX030)
Number analyzed (Participants) | 20
L/min | 0.293 [0.059 to 0.527]

7. Secondary Outcome: Change From Baseline of the Blood Flow for the Portal Vein (Study Part A (Serelaxin Treatment Group Only))
Description: A non-contrast magnetic resonance angiography (MRA) sequence was performed to acquire phase contrast blood flow measurements from vessels of interest such as the portal vein. The flow is the average flow over the cardiac cycle.
  Baseline blood flow measurements are measured at pre-dose (Day 1, 0 min post-treatment).
Time Frame: Baseline, 120 min post-infusion
Population: as for outcome 4
Measure: Mean (95% Confidence Interval); unit: L/min
Arm/Group | Part A: Serelaxin (RLX030)
Number analyzed (Participants) | 20
L/min | -0.091 [-0.204 to 0.023]

8. Secondary Outcome: Change From Baseline of the Portal Vein Pressure (PVP) (Study Part B)
Description: Portal vein pressure was measured at 15 min intervals (i.e. prior to and at 15, 30, 45, 60, 75, 90, 105, and 120 min of serelaxin infusion).
Time Frame: Baseline, 120 min post infusion
Population: For Part B of the study, full analysis set included all patients who received any amount of study treatment during the treatment period and had at least one post-baseline assessment during that period. Only patients with a value at both baseline and this time point are included.
Measure: Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Part B: Serelaxin (RLX030)
Number analyzed (Participants) | 6
mmHg | -3.7 [-8.8 to 1.4]

9. Secondary Outcome: Number of Patients With Total Adverse Events, Serious Adverse and Death as Assessment of Safety and Tolerability of Serelaxin
Description: This endpoint reports patients with any adverse event, serious adverse event and death for the serelaxin group of Part A and Part B of the study.
Time Frame: 4 weeks
Population: Safety assessment happened on full analysis set which included all patients who received any amount of study treatment during the treatment period and had at least one post-Baseline assessment during that period.
Measure: Number; unit: Patients
Arm/Group | Part A: Serelaxin (RLX030) | Part B: Serelaxin (RLX030)
Number analyzed (Participants) | 20 | 6
Patients
  Any adverse event | 3 | 3
  Serious Adverse Events | 1 | 2
  Death | 0 | 0

ADVERSE EVENTS:
Arm/Group | Part A: Serelaxin (RLX030) | Part A: Terlipressin Acetate | Part B: Serelaxin (RLX030)
Serious Adverse Events (participants affected / at risk) | 1/20 | 1/20 | 2/6
Other Adverse Events (participants affected / at risk) | 2/20 | 11/20 | 2/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: Serelaxin (RLX030) (N=20) | Part A: Terlipressin Acetate (N=20) | Part B: Serelaxin (RLX030) (N=6)
Ascites (Gastrointestinal disorders) | 1 | 0 | 0
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0
Hepatic encephalopathy (Nervous system disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: Serelaxin (RLX030) (N=20) | Part A: Terlipressin Acetate (N=20) | Part B: Serelaxin (RLX030) (N=6)
Abdominal pain (Gastrointestinal disorders) | 0 | 4 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 6 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 1 | 1 | 2
Electrocardiogram T wave biphasic (Investigations) | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.